CLINICAL TRIAL: NCT00263406
Title: Pathophysiological Mechanisms of Hepatopulmonary Influence in the Fontan Circulation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2002/055
Record Dates: First submitted 2005-12-04; First posted 2005-12-08 (Estimated); Last update posted 2007-12-28 (Estimated); Status verified 2007-12

CONDITIONS: Children With a Univentricular Heart Undergoing Surgery for Creation of a Fontan Circulation
MeSH Terms: interventions — Nuclear Receptor Subfamily 4, Group A, Member 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Administration of an ACE-inhibitor or not

SUMMARY:
Randomisation between postoperative administration of an ACE-inhibitor or not.

DETAILED DESCRIPTION:
Children that are undergoing elective surgery for the creation of a Fontan circulation will be randomised to postoperative administration of an ACE-inhibitor or not.

Determination of aldosteron, renine and ADH in serum preoperatively and 1h, 12h and 5 days postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* All consecutive children with a univentricular heart disease undergoing elective surgery for creation of a Fontan circulation
* Parents have agreed with the study after informed consent

Exclusion Criteria:

* Urgent / Emergent surgery
* Preoperative use of an ACE-inhibitor

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40
Dates: Start 2002-12; Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Duration of the pleural drainage in the first two postoperative weeks

CONTACTS AND LOCATIONS:
Overall Officials: Guy Van Nooten, MD, PhD, Principal Investigator — University Hospital, Ghent
Locations (1):
- University Hospital Ghent, Ghent, Belgium

REFERENCES:
- See also: Website of the University Hospital Ghent — http://www.uzgent.be